CLINICAL TRIAL: NCT04712760
Title: Congenital Hypothyroidism in Children With Eutopic Gland or Thyroid Hemiagenesis: Predictive Factors for Transient vs Permanent Hypothyroidism.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, RENARD Emeline, MD, Central Hospital, Nancy, France
Other Study IDs: 2020PI260
Record Dates: First submitted 2021-01-11; First posted 2021-01-15 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Congenital Hypothyroidism
Keywords: eutopic thyroid gland; transient hypothyroidism
MeSH Terms: conditions — Congenital Hypothyroidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transient congenital hypothyroidism: - children with congenital hypothyroidism who are no longer treated with Levothyroxine at an age of 3 years and 6 months
- Permanent congenital hypothyroidism: - children with congenital hypothyroidism who are still treated with Levothyroxine at an age of 3 years and 6 months

SUMMARY:
In France, the incidence of congenital hypothyroidism has increased significantly since the newborn screening program was introduced in 1978. The largest increase is seen in children with eutopic thyroid gland. More than one-third of children with eutopic gland have transient hypothyroidism. Clinical practice guidelines recommend to re-evaluate thyroid function in children with eutopic gland around the age of 3 years to determine whether hypothyroidism is transient or permanent. Up until today it is still difficult to determine early on whether hypothyroidism is transient or permanent in children with eutopic gland. Our aim is to identify one or more predictive factors for transient congenital hypothyroidism in children with eutopic gland or thyroid hemiagenesis.

ELIGIBILITY:
Inclusion Criteria:

* Children with congenital hypothyroidism
* Eutopic thyroid gland or thyroid hemiagenesis
* Born between 1996 and 2017
* Treated at the Nancy Regional and University Hospital
* Follow-up of at least 3,5 years.

Exclusion Criteria:

* Polymalformative syndrome
* Thyroid dysgenesis except for thyroid hemiagenesis

Max Age: 42 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with congenital hypothyroidism either detected by newborn screening or by a blood test done because of clinical suspicion of hypothyroidism, in Lorraine, between 1996 and 2017. All the patients with confirmed hypothyroidism underwent thyroid imaging. The children with eutopic gland and hemiagenesis are included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Identify one or more predictive factors for transient congenital hypothyroidism in children with eutopic gland or thyroid hemiagenesis. | 42 months

SECONDARY OUTCOMES:
Compare the dose of Levothyroxine between children with transient and permanent congenital hypothyroidism at 6 months, 1 year, 2 years and 3 years follow-up. | 6 months, 1 year, 2 years, 3 years
Assess the percentage of children with psychomotor impairment at the age of 3,5 years in both groups. | 42 months
Assess how many children have had a hearing evaluation in both groups (excluding the newborn hearing screening). | 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Emeline Renard, MD, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bontemps SH, Legagneur C, Gueant-Rodriguez RM, Remen T, Luc A, Renard E. Congenital hypothyroidism in children with eutopic gland or thyroid hemiagenesis: prognostic factors for transient vs. permanent hypothyroidism. J Pediatr Endocrinol Metab. 2023 Feb 20;36(4):353-363. doi: 10.1515/jpem-2022-0101. Print 2023 Apr 25. PMID 36798001